CLINICAL TRIAL: NCT05982769
Title: Molecular Mechanism of Exercise in Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-090
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Resistance Training; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endurance Arm (Experimental)
  Interventions: Behavioral: Endurance Training 3 times per week
- Resistance (Experimental)
  Interventions: Behavioral: Resistance Exercise
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Endurance Training 3 times per week — endurance training will be performed from home 3 times per week under the supervision of the research team.
  Arms: Endurance Arm
Behavioral: Resistance Exercise — resistance training will be performed from home 2 times per week under the supervision of the research team.
  Arms: Resistance
Behavioral: Standard of Care — continue usual activity
  Arms: Standard of Care

SUMMARY:
This study aims to investigate the effects of 12 weeks of resistance or endurance exercise on patients with cirrhosis. Cirrhotic patients are prone to muscle loss (sarcopenia) and ammonia build up due to liver dysfunction. The liver which in healthy patients is able to process ammonia through ureagenesis is unable to do so in cirrhosis and ammonia is taken up either by the brain causing confusion or the skeletal muscle causing muscle loss or sarcopenia. Primary sarcopenia occurs in older individuals and can be mitigated by exercise. Secondary sarcopenia occurs in response to disease such as cancer, chronic kidney disease, multiple sclerosis, and cirrhosis of all etiologies. Resistance exercise is an excellent stimulator for muscle protein synthesis and is widely used to build muscle mass and strength but has little benefit to cardiovascular function. Endurance exercise has shown to be safe in cirrhosis however there is no set prescription for cirrhosis as there is for other disease. Endurance exercise is known to promote improved cardiovascular health, improve fatigue, and generates less ammonia build up than resistance exercise. In patients with low muscle mass it is possible that endurance exercise alone will be enough to improve muscle mass. There have been few studies on exercise and cirrhosis, those that exist have shown benefits with endurance exercise. However there are even more limited studies on resistance exercise and few to no studies on the molecular mechanisms behind exercise in cirrhosis. Study visits are described fully in the protocol and consent form. After passing a screening visit patients will undergo a maximal exercise/fitness test (pre-baseline test) and other body composition measurements. After the screening and pre-baseline visit randomization will occur (2:2:1 endurance, resistance, or SOC) arrangements will be made to have the appropriate exercise equipment given to patients. Once the exercise equipment has arrived a baseline study visit will occur. After the baseline visit the endurance exercise group will cycle 3 days per week for 60 minutes under the supervision of the study team. The resistance exercise group will perform a whole body resistance workout 2 days per week for approximately 60 minutes under the supervision of a study team member.

Patients in all groups will have the fitness test repeated at weeks 4, 8 and 12. After the 12 weeks of exercise the baseline visits will be repeated and after 2 weeks patients will complete one final fitness test to examine the effects of de-training.

ELIGIBILITY:
Inclusion

* Adult patients age 21-65 years of both genders
* Diagnosis of cirrhosis by either liver biopsy, clinical, biochemical or imaging criteria
* Child's score 5-10
* Model for End Stage Liver Disease (MELD) score less than 21
* Abstinence from alcohol and/or other recreational drugs for at least 6 months
* Absence of concurrent illnesses (renal, cardiac, pulmonary, cerebrovascular, malignancy) or medication (anabolic steroids, corticosteroids) intake that affect skeletal muscle mass, diabetes mellitus (avoid altered muscle protein metabolism), or use of anticoagulants.
* abdominal or liver CT scan within 1 year of enrollment for stratification Exclusion
* Active alcohol consumption within 6 weeks of enrollment
* Pedal edema (grade 2) above the ankle will be excluded to avoid complications of the muscle biopsy.
* Liver transplant
* Active Malignancy
* Recent GI bleed (4 weeks)
* Hepatic Encephalopathy within previous 6 months
* Grade 2 or greater active esophageal varices
* Active infection
* Large Ascites as defined by clinical imaging
* Advanced disease cardiac or pulmonary disease
* Use of medications affecting muscle protein turnover including corticosteroids or medications used to prevent clotting
* Clinical lab values that indicate potential poor clotting as determined by the PI
* Inability to obtain informed consent; judged likely to be unable to perform exercise or unlikely to complete the study in the opinion of the investigators
* End stage kidney disease as determined by glomerular filtration rate (eGFR) < 15 ml/min/1.73m2 or dialysis
* Patients who in the opinion of the PI are unsafe for exercise (failure to pass stress test)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in muscle mass over time | day 0 and day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No